CLINICAL TRIAL: NCT06732401
Title: A Randomized Phase III Trial of Checkpoint Blockade in Lung Cancer Patients in the Adjuvant Setting Based on Pathologic Response Following Neoadjuvant Therapy (CLEAR)
Brief Title: Testing the Addition of AZD6738 (Ceralasertib) to Immunotherapy to Increase Time Without Cancer for Patients With Non-Small Cell Lung Cancer
Status: Suspended | Phase: Phase 3 | Type: Interventional
Why Stopped: Other - Per CTEP request due to new data with agent
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2024-10081; NCI-2024-10081 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); EA5231 (Other: ECOG-ACRIN Cancer Research Group); EA5231 (Other: CTEP); U10CA180820 (NIH)
Record Dates: First submitted 2024-12-12; First posted 2024-12-13 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-01

CONDITIONS: Lung Non-Small Cell Carcinoma; Stage II Lung Cancer AJCC v8; Stage IIIA Lung Cancer AJCC v8; Stage IIIB Lung Cancer AJCC v8
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Lung Neoplasms | interventions — Specimen Handling; ceralasertib; durvalumab; Immunoglobulin G; Disulfides

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm A (Durvalumab) (Active Comparator): Starting 4-12 weeks after surgery, patients receive durvalumab IV over 60 minutes on day 1 of each cycle. Cycles repeat every 28 days for 12 cycles in the absence of disease progression or unacceptable toxicity. Patients undergo CT scan and blood sample collection throughout the study and may undergo echocardiography as clinically indicated.
  Interventions: Procedure: Biospecimen Collection; Procedure: Computed Tomography; Biological: Durvalumab; Procedure: Echocardiography Test
- Arm B (Durvalumab and AZD6738) (Experimental): Starting 4-12 weeks after surgery, patients receive AZD6738 PO BID on days 1-7 and durvalumab IV over 60 minutes on day 8 of each cycle. Cycles repeat every 28 days for 12 cycles in the absence of disease progression or unacceptable toxicity. Patients undergo CT scan and blood sample collection throughout the study and may undergo echocardiography as clinically indicated.
  Interventions: Procedure: Biospecimen Collection; Drug: Ceralasertib; Procedure: Computed Tomography; Biological: Durvalumab; Procedure: Echocardiography Test

INTERVENTIONS:
Procedure: Biospecimen Collection — Undergo blood sample collection
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Drug: Ceralasertib — Given PO
  Other Names: AZD6738
  Arms: Arm B (Durvalumab and AZD6738)
Procedure: Computed Tomography — Undergo CT scan
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized axial tomography (procedure); Computerized Tomography; Computerized Tomography (CT) scan; CT; CT Scan; Diagnostic CAT Scan; Diagnostic CAT Scan Service Type; tomography
Biological: Durvalumab — Given IV
  Other Names: Imfinzi; Immunoglobulin G1, Anti-(Human Protein B7-H1) (Human Monoclonal MEDI4736 Heavy Chain), Disulfide with Human Monoclonal MEDI4736 Kappa-chain, Dimer; MEDI 4736; MEDI-4736; MEDI4736
Procedure: Echocardiography Test — Undergo echocardiography
  Other Names: EC; Echocardiography

SUMMARY:
This phase III trial compares the effect of adding AZD6738 to durvalumab versus durvalumab alone to increase time without cancer in patients with non-small cell lung cancer, following treatment with chemotherapy and surgery. AZD6738 may stop the growth of tumor cells and may kill them by blocking some of the enzymes needed for cell growth. Durvalumab is a monoclonal antibody that may interfere with the ability of tumor cells to grow and spread. A monoclonal antibody is a type of protein that can bind to certain targets in the body, such as molecules that cause the body to make an immune response (antigens). Adding AZD6738 to durvalumab may increase time without cancer in patients with non-small cell lung cancer, following treatment with chemotherapy and surgery.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To assess for improvement in disease free survival (DFS) in patients who do not achieve pathologic complete response (pCR) following neoadjuvant therapy and patients who receive adjuvant combination immunotherapy with durvalumab and AZD6738 (ceralasertib) compared to those who receive monotherapy with durvalumab.

SECONDARY OBJECTIVE:

I. To evaluate any difference in overall survival (OS) with patients who receive durvalumab and AZD6738 (ceralasertib) compared to those who receive monotherapy with durvalumab.

EXPLORATORY OBJECTIVES:

I. To evaluate any difference in disease free survival (DFS) with patients who receive durvalumab and AZD6738 (ceralasertib) compared to those who receive monotherapy with durvalumab according to PD-L1, stage, prior immune checkpoint inhibitor (ICI) type, and histology.

II. To evaluate any difference in overall survival (OS) with patients who receive durvalumab and AZD6738 (ceralasertib) compared to those who receive monotherapy with durvalumab according to PD-L1, stage, prior ICI type, and histology.

CORRELATIVE OBJECTIVE:

I. To perform correlative analyses on tissue and blood biospecimens collected within this trial.

OUTLINE: Patients are randomized to 1 of 2 arms.

ARM A: Starting 4-12 weeks after surgery, patients receive durvalumab intravenously (IV) over 60 minutes on day 1 of each cycle. Cycles repeat every 28 days for 12 cycles in the absence of disease progression or unacceptable toxicity. Patients undergo computed tomography (CT) scan and blood sample collection throughout the study and may undergo echocardiography as clinically indicated.

ARM B: Starting 4-12 weeks after surgery, patients receive AZD6738 orally (PO) twice daily (BID) on days 1-7 and durvalumab IV over 60 minutes on day 8 of each cycle. Cycles repeat every 28 days for 12 cycles in the absence of disease progression or unacceptable toxicity. Patients undergo CT scan and blood sample collection throughout the study and may undergo echocardiography as clinically indicated.

After completion of study treatment, patients are followed up every 12 weeks for 2 years then every 24 weeks until year 5 then every 12 months until 10 years from randomization.

ELIGIBILITY:
Inclusion Criteria:

* STEP 0: Patient must be >= 18 years of age
* STEP 0: Patient must have stage II to select stage IIIB (N2 but excluding N3) non-small cell lung cancer (NSCLC) of any histology using International Association for the Study of Lung Cancer (IASLC) 8th edition. Stage is assessed at time of initiating pre-operative chemo-immunotherapy
* STEP 0: Patient must fall into one of the following categories:

  * Planning to undergo, be currently undergoing, or recently completed any standard of care neoadjuvant chemo-immunotherapy with plans to undergo surgical resection
  * Recently completed any standard of care neoadjuvant chemo-immunotherapy AND completed surgical resection and are awaiting pCR status.
  * Recently completed any standard of care neoadjuvant chemo-immunotherapy AND completed surgical resection with confirmed non-path complete response (CR) status.

NOTES:

* Patient must have completed at least 3 cycles of neoadjuvant chemo-immunotherapy before surgery in order to be eligible for Step 1 randomization.
* Patients who have completed their surgical resection prior to enrollment in step 0 registration must have their surgery date within a window that will allow initiation of EA5231 treatment (cycle 1 day 1) to commence within 4-12 weeks following surgery

  * STEP 1: EA5231 CLEAR randomization for patients without a pCR post-surgery. Patient's with pCR after surgery will be offered to enroll in the SWOG study S2414 INSIGHT instead
  * STEP 1: Patient must have completed R0 resection after standard of care neoadjuvant chemo-immunotherapy (minimum three cycles completed) for stage II to select stage IIIB (N2 but excluding N3) non-small cell lung cancer (NSCLC) of any histology using IASLC 8th Edition
  * STEP 1: Patient must have non-pathological CR status post-surgery. The pathological CR/non-pathological CR status will be determined by local pathology using IASLC criteria and using the surgical sample tissue
  * STEP 1: Patient must have an Eastern Cooperative Oncology Group (ECOG) performance status of 0 - ≤ 2 (or Karnofsky ≥ 60%)
  * STEP 1: Patient must not have any known EGFR or ALK genetic alterations. Mutation negative status will be determined per local institutional practices and consistent with National Comprehensive Cancer Network (NCCN) guidelines
  * STEP 1: Patient must have undergone a chest CT after surgery and within 28 days prior to step 1 randomization
  * STEP 1: Patient must have recovered from clinically significant adverse events of their most recent therapy/intervention prior to step 1 randomization
  * STEP 1: Patient must not have experienced a toxicity that led to the permanent discontinuation of prior immunotherapy
  * STEP 1: Patient must not be receiving ongoing steroids at a dose of prednisone 10 mg or higher (or equivalent) at the time of step 1 randomization. Steroids as premedication for hypersensitivity reactions (e.g., CT scan premedication) are allowed. Intranasal, inhaled, topical steroids, or local steroid injections (e.g., intra articular injection) are allowed
  * STEP 1: Patient must not have received or have a plan to receive post-operative radiation therapy (PORT)
  * STEP 1: Patient must not have a history of treatment-related pneumonitis requiring ongoing steroids or supplemental oxygen use
  * STEP 1: Patient must not have a history of interstitial lung disease (ILD)
  * STEP 1: Patient must not have diagnosis of ataxia telangiectasia
  * STEP 1: Patient must not have history of active primary immunodeficiency
  * STEP 1: Patient must not have history of allogenic organ transplantation
  * STEP 1: Patient must have body weight > 30 kg
  * STEP 1: Patient must not be pregnant or breast-feeding due to the potential harm to an unborn fetus and possible risk for adverse events in nursing infants with the treatment regimens being used. All patients of childbearing potential must have a blood test or urine study within 14 days prior to Step 1 randomization to rule out pregnancy. A patient of childbearing potential is defined as anyone, regardless of whether they have undergone tubal ligation, who meets the following criteria:
* Has achieved menarche at some point
* Has not undergone a hysterectomy or bilateral oophorectomy
* Has not been naturally postmenopausal (amenorrhea following cancer therapy does not rule out childbearing potential) for at least 24 consecutive months (i.e., has had menses at any time in the preceding 24 consecutive months)

  * STEP 1: Patient must not expect to conceive or father children by using highly accepted and effective method(s) of contraception or by abstaining from sexual intercourse for the duration of their participation in the study. Patients of childbearing potential must use at least 1 highly effective method of contraception in addition to a condom and continue to use it throughout their time on protocol treatment. Male patients must use a condom plus spermicide throughout their time on while on protocol treatment. In addition, all patients must continue contraception use for at least 6 months after the last dose of protocol treatment. Patients must also not breastfeed while on protocol treatment and for at least 6 months after the last dose of protocol treatment. Patients must not donate sperm while on protocol treatment and for 6 months after the last dose of protocol treatment
  * STEP 1: Patient must not donate blood while on protocol treatment
  * STEP 1: Patient must have the ability to understand and the willingness to sign a written informed consent document. Patients with impaired decision-making capacity (IDMC) who have a legally authorized representative (LAR) or caregiver and/or family member available will also be considered eligible
  * STEP 1: Leukocytes ≥ 3,000/mcL (these labs must be obtained ≤ 28 days prior to step 1 randomization)
  * STEP 1: Hemoglobin ≥ 9.0 g/dL (these labs must be obtained ≤ 28 days prior to step 1 randomization)
  * STEP 1: Absolute neutrophil count (ANC) ≥ 1,500/mcL (these labs must be obtained ≤ 28 days prior to step 1 randomization)
  * STEP 1: Platelets ≥ 100,000/mcL (these labs must be obtained ≤ 28 days prior to step 1 randomization)
  * STEP 1: Total bilirubin ≤ institutional upper limit of normal (ULN) (these labs must be obtained ≤ 28 days prior to step 1 randomization)
  * STEP 1: Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT]) and alanine aminotransferase (ALT) (serum glutamic pyruvic transaminase [SGPT]) ≤ 3.0 × institutional ULN (these labs must be obtained ≤ 28 days prior to step 1 randomization)
  * STEP 1: Creatinine clearance ≥ 50 mL/min (estimated using Cockcroft-Gault method or measured) (these labs must be obtained ≤ 28 days prior to step 1 randomization)
  * STEP 1: Human immunodeficiency virus (HIV)-infected patients on effective anti-retroviral therapy with undetectable viral load within 6 months of step 1 randomization are eligible for this trial
  * STEP 1: For patients with known chronic hepatitis B virus (HBV) infection, the HBV viral load must be undetectable on suppressive therapy, if indicated
  * STEP 1: Patients with a history of hepatitis C virus (HCV) infection must have been treated and cured. For patients with HCV infection who are currently on treatment, they are eligible if they have an undetectable HCV viral load
  * STEP 1: Patients with a prior or concurrent malignancy whose natural history or treatment does not have the potential to interfere with the safety or efficacy assessment of the investigational regimen are eligible for this trial
  * STEP 1: Patients with known history or current symptoms of cardiac disease, or history of treatment with cardiotoxic agents, should have a clinical risk assessment of cardiac function using the New York Heart Association Functional Classification. To be eligible for this trial, patients should be class 2B or better
  * STEP 1: Patient must not have received live attenuated vaccine within 30 days prior to the step 1 randomization, while on protocol treatment and within 30 days after the last dose of durvalumab

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 630 (Estimated)
Dates: Start 2025-08-07 (Actual); Primary Completion 2028-06-30 (Estimated); Study Completion 2028-06-30 (Estimated)

PRIMARY OUTCOMES:
Disease free survival (DFS) | From randomization to the earliest event defined as the first recurrence of non-small cell lung cancer (NSCLC), any new lung cancer or death, up to 10 years
  Will estimate DFS distributions using the Kaplan-Meier method and employ Cox proportional hazards models to estimate the treatment hazard ratios. The comparison of DFS will use a logrank test stratified on the randomization stratification factors with a one-sided type I error rate of 2.5%. Other comparisons of groups will be made using the logrank test and Cox modeling. Point estimates will be accompanied by the corresponding two-sided 95% confidence intervals.

SECONDARY OUTCOMES:
Overall survival (OS) | From randomization to death from any cause, up to 10 years
  Will estimate OS distributions using the Kaplan-Meier method and employ Cox proportional hazards models to estimate the treatment hazard ratios. The comparison of OS will use a logrank test stratified on the randomization stratification factors with a one-sided type I error rate of 2.5%. Other comparisons of groups will be made using the logrank test and Cox modeling. Point estimates will be accompanied by the corresponding two-sided 95% confidence intervals.
Incidence of adverse events | Up to 10 years
  Toxicity will be assessed by summaries by Common Terminology Criteria for Adverse Event grade.

OTHER OUTCOMES:
Estimates of treatment effect by sex | Up to 10 years
  Estimates of DFS and the corresponding 95% confidence intervals (CIs) by sex.
Estimates of treatment effect by race | Up to 10 years
  Estimates of DFS and the corresponding 95% CIs by race.
Estimates of treatment effect by ethnicity | Up to 10 years
  Estimates of DFS and the corresponding 95% CIs by ethnicity.
DFS according to PD-L1 status | Up to 10 years
  Will be compared between treatment arms using the logrank test and Cox modeling.
DFS according to stage | Up to 10 years
  Will be compared between treatment arms using the logrank test and Cox modeling.
DFS according to prior immune checkpoint inhibitor (ICI) type | Up to 10 years
  Will be compared between treatment arms using the logrank test and Cox modeling.
DFS according to histology | Up to 10 years
  Will be compared between treatment arms using the logrank test and Cox modeling.
OS according to PD-L1 status | Up to 10 years
  Will be compared between treatment arms using the logrank test and Cox modeling.
OS according to stage | Up to 10 years
  Will be compared between treatment arms using the logrank test and Cox modeling.
OS according to prior ICI type | Up to 10 years
  Will be compared between treatment arms using the logrank test and Cox modeling.
OS according to histology | Up to 10 years
  Will be compared between treatment arms using the logrank test and Cox modeling.
Correlative analyses on tissue, blood, and stool biospecimens | Up to 10 years

CONTACTS AND LOCATIONS:
Overall Officials: Dwight H Owen, Principal Investigator — ECOG-ACRIN Cancer Research Group
Locations (193):
- United States (193):
  - NEA Baptist Memorial Hospital and Fowler Family Cancer Center - Jonesboro, Jonesboro, Arkansas
  - Tower Cancer Research Foundation, Beverly Hills, California
  - Cedars Sinai Medical Center, Los Angeles, California
  - Cedars-Sinai Cancer - Tarzana, Tarzana, California
  - Torrance Memorial Physician Network - Cancer Care, Torrance, California
  - Hartford Hospital, Hartford, Connecticut
  - Midstate Medical Center, Meriden, Connecticut
  - The Hospital of Central Connecticut, New Britain, Connecticut
  - Beebe South Coastal Health Campus, Millville, Delaware
  - Helen F Graham Cancer Center, Newark, Delaware
  - Medical Oncology Hematology Consultants PA, Newark, Delaware
  - Beebe Health Campus, Rehoboth Beach, Delaware
  - MedStar Georgetown University Hospital, Washington D.C., District of Columbia
  - MedStar Washington Hospital Center, Washington D.C., District of Columbia
  - Emory University Hospital Midtown, Atlanta, Georgia
  - Emory University Hospital/Winship Cancer Institute, Atlanta, Georgia
  - Emory Saint Joseph's Hospital, Atlanta, Georgia
  - Emory Decatur Hospital, Decatur, Georgia
  - Emory Johns Creek Hospital, Johns Creek, Georgia
  - Saint Luke's Cancer Institute - Boise, Boise, Idaho
  - Kootenai Health - Coeur d'Alene, Coeur d'Alene, Idaho
  - Saint Luke's Cancer Institute - Fruitland, Fruitland, Idaho
  - Saint Luke's Cancer Institute - Meridian, Meridian, Idaho
  - Saint Alphonsus Cancer Care Center-Nampa, Nampa, Idaho
  - Saint Luke's Cancer Institute - Nampa, Nampa, Idaho
  - Kootenai Clinic Cancer Services - Post Falls, Post Falls, Idaho
  - Kootenai Clinic Cancer Services - Sandpoint, Sandpoint, Idaho
  - Illinois CancerCare-Bloomington, Bloomington, Illinois
  - Illinois CancerCare-Canton, Canton, Illinois
  - Illinois CancerCare-Carthage, Carthage, Illinois
  - Northwestern University, Chicago, Illinois
  - Cancer Care Specialists of Illinois - Decatur, Decatur, Illinois
  - Decatur Memorial Hospital, Decatur, Illinois
  - Northwestern Medicine Cancer Center Kishwaukee, DeKalb, Illinois
  - Illinois CancerCare-Dixon, Dixon, Illinois
  - Crossroads Cancer Center, Effingham, Illinois
  - Illinois CancerCare-Eureka, Eureka, Illinois
  - Illinois CancerCare-Galesburg, Galesburg, Illinois
  - Northwestern Medicine Cancer Center Delnor, Geneva, Illinois
  - Northwestern Medicine Glenview Outpatient Center, Glenview, Illinois
  - Northwestern Medicine Grayslake Outpatient Center, Grayslake, Illinois
  - Illinois CancerCare-Kewanee Clinic, Kewanee, Illinois
  - Northwestern Medicine Lake Forest Hospital, Lake Forest, Illinois
  - Illinois CancerCare-Macomb, Macomb, Illinois
  - Loyola University Medical Center, Maywood, Illinois
  - Cancer Care Center of O'Fallon, O'Fallon, Illinois
  - HSHS Saint Elizabeth's Hospital, O'Fallon, Illinois
  - Northwestern Medicine Oak Brook, Oak Brook, Illinois
  - Northwestern Medicine Orland Park, Orland Park, Illinois
  - Illinois CancerCare-Ottawa Clinic, Ottawa, Illinois
  - Illinois CancerCare-Pekin, Pekin, Illinois
  - Illinois CancerCare-Peoria, Peoria, Illinois
  - Illinois CancerCare-Peru, Peru, Illinois
  - Illinois CancerCare-Princeton, Princeton, Illinois
  - Southern Illinois University School of Medicine, Springfield, Illinois
  - Springfield Clinic, Springfield, Illinois
  - Springfield Memorial Hospital, Springfield, Illinois
  - Northwestern Medicine Cancer Center Warrenville, Warrenville, Illinois
  - Illinois CancerCare - Washington, Washington, Illinois
  - Indiana University/Melvin and Bren Simon Cancer Center, Indianapolis, Indiana
  - Cancer Center of Kansas - El Dorado, El Dorado, Kansas
  - Lawrence Memorial Hospital, Lawrence, Kansas
  - Cancer Center of Kansas - Newton, Newton, Kansas
  - The University of Kansas Cancer Center - Olathe, Olathe, Kansas
  - Salina Regional Health Center, Salina, Kansas
  - University of Kansas Health System Saint Francis Campus, Topeka, Kansas
  - Cancer Center of Kansas - Wellington, Wellington, Kansas
  - Cancer Center of Kansas-Wichita Medical Arts Tower, Wichita, Kansas
  - Ascension Via Christi Hospitals Wichita, Wichita, Kansas
  - Cancer Center of Kansas - Wichita, Wichita, Kansas
  - Cancer Center of Kansas - Winfield, Winfield, Kansas
  - University of Maryland/Greenebaum Cancer Center, Baltimore, Maryland
  - UM Baltimore Washington Medical Center/Tate Cancer Center, Glen Burnie, Maryland
  - Beverly Hospital, Beverly, Massachusetts
  - Lahey Hospital and Medical Center, Burlington, Massachusetts
  - Addison Gilbert Hospital, Gloucester, Massachusetts
  - Lahey Medical Center-Peabody, Peabody, Massachusetts
  - Baystate Medical Center, Springfield, Massachusetts
  - Bronson Battle Creek, Battle Creek, Michigan
  - Trinity Health IHA Medical Group Hematology Oncology - Brighton, Brighton, Michigan
  - Trinity Health IHA Medical Group Hematology Oncology - Canton, Canton, Michigan
  - Trinity Health IHA Medical Group Hematology Oncology - Chelsea Hospital, Chelsea, Michigan
  - Cancer Hematology Centers - Flint, Flint, Michigan
  - Genesee Hematology Oncology PC, Flint, Michigan
  - Genesys Hurley Cancer Institute, Flint, Michigan
  - Hurley Medical Center, Flint, Michigan
  - Corewell Health Grand Rapids Hospitals - Butterworth Hospital, Grand Rapids, Michigan
  - Trinity Health Grand Rapids Hospital, Grand Rapids, Michigan
  - Bronson Methodist Hospital, Kalamazoo, Michigan
  - West Michigan Cancer Center, Kalamazoo, Michigan
  - University of Michigan Health - Sparrow Lansing, Lansing, Michigan
  - Trinity Health Saint Mary Mercy Livonia Hospital, Livonia, Michigan
  - Trinity Health Muskegon Hospital, Muskegon, Michigan
  - Corewell Health Lakeland Hospitals - Niles Hospital, Niles, Michigan
  - Cancer and Hematology Centers of Western Michigan - Norton Shores, Norton Shores, Michigan
  - Trinity Health Saint Joseph Mercy Oakland Hospital, Pontiac, Michigan
  - Corewell Health Reed City Hospital, Reed City, Michigan
  - Corewell Health Lakeland Hospitals - Marie Yeager Cancer Center, Saint Joseph, Michigan
  - Corewell Health Lakeland Hospitals - Saint Joseph Hospital, Saint Joseph, Michigan
  - Munson Medical Center, Traverse City, Michigan
  - University of Michigan Health - West, Wyoming, Michigan
  - Trinity Health IHA Medical Group Hematology Oncology Ann Arbor Campus, Ypsilanti, Michigan
  - Essentia Health Saint Joseph's Medical Center, Brainerd, Minnesota
  - Mercy Hospital, Coon Rapids, Minnesota
  - Essentia Health - Deer River Clinic, Deer River, Minnesota
  - Essentia Health Cancer Center, Duluth, Minnesota
  - Fairview Southdale Hospital, Edina, Minnesota
  - Essentia Health Hibbing Clinic, Hibbing, Minnesota
  - Abbott-Northwestern Hospital, Minneapolis, Minnesota
  - Minneapolis VA Medical Center, Minneapolis, Minnesota
  - Park Nicollet Clinic - Saint Louis Park, Saint Louis Park, Minnesota
  - Regions Hospital, Saint Paul, Minnesota
  - United Hospital, Saint Paul, Minnesota
  - Essentia Health Sandstone, Sandstone, Minnesota
  - Essentia Health Virginia Clinic, Virginia, Minnesota
  - Baptist Memorial Hospital and Cancer Center-Golden Triangle, Columbus, Mississippi
  - Baptist Cancer Center-Grenada, Grenada, Mississippi
  - Baptist Memorial Hospital and Cancer Center-Union County, New Albany, Mississippi
  - Baptist Memorial Hospital and Cancer Center-Oxford, Oxford, Mississippi
  - Baptist Memorial Hospital and Cancer Center-Desoto, Southhaven, Mississippi
  - Saint Francis Medical Center, Cape Girardeau, Missouri
  - Parkland Health Center - Farmington, Farmington, Missouri
  - Sainte Genevieve County Memorial Hospital, Sainte Genevieve, Missouri
  - Mercy Hospital South, St Louis, Missouri
  - Missouri Baptist Medical Center, St Louis, Missouri
  - Missouri Baptist Sullivan Hospital, Sullivan, Missouri
  - BJC Outpatient Center at Sunset Hills, Sunset Hills, Missouri
  - Community Hospital of Anaconda, Anaconda, Montana
  - Billings Clinic Cancer Center, Billings, Montana
  - Saint Vincent Frontier Cancer Center, Billings, Montana
  - Bozeman Health Deaconess Hospital, Bozeman, Montana
  - Benefis Sletten Cancer Institute, Great Falls, Montana
  - Community Medical Center, Missoula, Montana
  - New Hampshire Oncology Hematology PA-Concord, Concord, New Hampshire
  - Solinsky Center for Cancer Care, Manchester, New Hampshire
  - Hunterdon Medical Center, Flemington, New Jersey
  - Glens Falls Hospital, Glens Falls, New York
  - Montefiore Medical Center-Einstein Campus, The Bronx, New York
  - FirstHealth of the Carolinas-Moore Regional Hospital, Pinehurst, North Carolina
  - Essentia Health Cancer Center-South University Clinic, Fargo, North Dakota
  - Aultman Health Foundation, Canton, Ohio
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Providence Newberg Medical Center, Newberg, Oregon
  - Providence Willamette Falls Medical Center, Oregon City, Oregon
  - Providence Portland Medical Center, Portland, Oregon
  - Providence Saint Vincent Medical Center, Portland, Oregon
  - Oregon Health and Science University, Portland, Oregon
  - Lehigh Valley Hospital-Cedar Crest, Allentown, Pennsylvania
  - Lehigh Valley Hospital - Muhlenberg, Bethlehem, Pennsylvania
  - Bryn Mawr Hospital, Bryn Mawr, Pennsylvania
  - Pocono Medical Center, East Stroudsburg, Pennsylvania
  - UPMC Hillman Cancer Center Erie, Erie, Pennsylvania
  - UPMC Cancer Centers - Arnold Palmer Pavilion, Greensburg, Pennsylvania
  - UPMC Pinnacle Cancer Center/Community Osteopathic Campus, Harrisburg, Pennsylvania
  - Lehigh Valley Hospital-Hazleton, Hazleton, Pennsylvania
  - UPMC Hillman Cancer Center at Rocco And Nancy Ortenzio Cancer Pavilion, Mechanicsburg, Pennsylvania
  - Riddle Memorial Hospital, Media, Pennsylvania
  - UPMC Hillman Cancer Center - Monroeville, Monroeville, Pennsylvania
  - Paoli Memorial Hospital, Paoli, Pennsylvania
  - University of Pennsylvania/Abramson Cancer Center, Philadelphia, Pennsylvania
  - University of Pittsburgh Cancer Institute (UPCI), Pittsburgh, Pennsylvania
  - UPMC-Saint Clair Hospital Cancer Center, Pittsburgh, Pennsylvania
  - Reading Hospital, West Reading, Pennsylvania
  - Lankenau Medical Center, Wynnewood, Pennsylvania
  - Tidelands Georgetown Memorial Hospital, Georgetown, South Carolina
  - Baptist Memorial Hospital and Cancer Center-Collierville, Collierville, Tennessee
  - Baptist Memorial Hospital and Cancer Center-Memphis, Memphis, Tennessee
  - Vanderbilt University/Ingram Cancer Center, Nashville, Tennessee
  - University of Virginia Cancer Center, Charlottesville, Virginia
  - Hematology Oncology Associates of Fredericksburg Inc, Fredericksburg, Virginia
  - Virginia Cancer Institute, Richmond, Virginia
  - VCU Massey Cancer Center at Stony Point, Richmond, Virginia
  - VCU Massey Comprehensive Cancer Center, Richmond, Virginia
  - VCU Community Memorial Health Center, South Hill, Virginia
  - Edwards Comprehensive Cancer Center, Huntington, West Virginia
  - West Virginia University Healthcare, Morgantown, West Virginia
  - Camden Clark Medical Center, Parkersburg, West Virginia
  - Langlade Hospital and Cancer Center, Antigo, Wisconsin
  - ThedaCare Regional Cancer Center, Appleton, Wisconsin
  - Duluth Clinic Ashland, Ashland, Wisconsin
  - Essentia Health-Hayward Clinic, Hayward, Wisconsin
  - Gundersen Lutheran Medical Center, La Crosse, Wisconsin
  - Aspirus Medford Hospital, Medford, Wisconsin
  - ProHealth D N Greenwald Center, Mukwonago, Wisconsin
  - ProHealth Oconomowoc Memorial Hospital, Oconomowoc, Wisconsin
  - Aspirus Cancer Care - James Beck Cancer Center, Rhinelander, Wisconsin
  - Essentia Health-Spooner Clinic, Spooner, Wisconsin
  - Aspirus Cancer Care - Stevens Point, Stevens Point, Wisconsin
  - Essentia Health Saint Mary's Hospital - Superior, Superior, Wisconsin
  - UW Cancer Center at ProHealth Care, Waukesha, Wisconsin
  - Aspirus Regional Cancer Center, Wausau, Wisconsin
  - Aspirus Cancer Care - Wisconsin Rapids, Wisconsin Rapids, Wisconsin

IPD SHARING:
Plan to Share IPD: Yes
NCI is committed to sharing data in accordance with NIH policy. For more details on how clinical trial data is shared, access the link to the NIH data sharing policy page.
URL: https://grants.nih.gov/policy/sharing.htm